CLINICAL TRIAL: NCT05199571
Title: A 12-month, Open-label, Prospective, Multicenter, Interventional, Single-arm Study Assessing the Efficacy and Safety of Ofatumumab 20 mg Subcutaneous (s.c.) Injection in Relapsing Multiple Sclerosis (RMS) Patients in China
Brief Title: Study of Efficacy and Safety of Ofatumumab in Relapsing Multiple Sclerosis (RMS) Patients in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157G2402
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing multiple sclerosis; open-label; interventional; efficacy and safety; ofatumumab; China; adult; OMB157
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ofatumumab (Experimental): Ofatumumab 20 mg subcutaneous injections at Week 0, 1, 2 and monthly thereafter starting at Week 4
  Interventions: Biological: Ofatumumab

INTERVENTIONS:
Biological: Ofatumumab — Solution for injection in an autoinjector (pre-filled pen) containing 20 mg ofatumumab
  Other Names: OMB157

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of ofatumumab s.c. in adult participants with relapsing multiple sclerosis (RMS) in China.

DETAILED DESCRIPTION:
This study consisted of three periods, Screening (up to 30 days), Treatment (12 months) and Post-treatment follow-up (6 months). It was an open-label single-arm study so all participants received the study drug. The first dose was administered in the clinic and the remaining doses were administered at home. The doses were administered at Baseline/Week 0, Week 1, Week 2, and followed by subsequent monthly dosing starting at Week 4.

Participants were required to come into the clinic for one screening visit, and 5 visits during the Treatment period for clinical evaluation and lab tests. Participants who completed the 12-month treatment had Post treatment Follow-Up visits at End of Study plus 3 months (EOS + 3M) and EOS + 6M, unless the participants decided to continue with commercially available ofatumumab treatment outside of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese aged 18-55 years (inclusive) at their enrollment of the study (signing the study consent form).
* Clinical definite diagnosis of RMS according to the 2017 Revised McDonald criteria (Thompson et al 2018, and the documentation prior to their enrollment to the study (signing the study consent form) of:

  * Two documented relapses during the past 2 years, or
  * One documented relapse during the last year, or
  * A positive Gd-enhancing MRI scan during the year prior to Screening. Note: Screening MRI scan may be used if no positive Gd-enhancing scan exists from prior year.
* Disability status with an EDSS score of 0 - 5.5 (inclusive) at Screening.
* Neurologically stable within 1 month prior to both Screening and Baseline (including no MS relapse in this period).

Exclusion Criteria:

* Participants with primary progressive MS (PPMS) or secondary progressive MS (SPMS) without disease activity
* Participants meeting criteria for neuromyelitis optica spectrum disorder (NMOSD)
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless using effective methods of contraception while taking study treatment and for at least 6 months after stopping medication
* Participants with an active chronic disease of the immune system other than MS
* Participants with neurological findings consistent with PML or confirmed PML
* Participants with active hepatitis B disease
* Participants with active systemic infections (including but not limited to active COVID-19 infection) or known to have AIDS or to test positive for HIV antibody at Screening
* Participants at high risk of developing or having reactivation of syphilis or tuberculosis
* Have received any live or live-attenuated vaccines within four weeks prior to first study drug administration
* Have been treated with medications as specified or within timeframes specified in the protocol
* Any other disease or condition that could interfere with participation in the study according to the study protocol, or with the ability of the participants to cooperate and comply with the study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Novartis Investigative Site, Lanzhou, Gansu
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shenzhen
  - Novartis Investigative Site, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=3031

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 19 sites in China
Pre-assignment Details: There were up to 30 days of screening period (day -30 to -1) before first treatment (day 1).
Period: Treatment period
Arm/Group | Ofatumumab
Started | 99
Completed | 95
Not Completed | 4
Not completed — Participant decision | 3
Not completed — Physician Decision | 1
Period: Post-treatment follow up period
Arm/Group | Ofatumumab
Started | 29
Completed | 26
Not Completed | 3
Not completed — Participant decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.98)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years | 0
  18 to 30 years | 46
  31 to 40 years | 38
  41 to 55 years | 15
  > 55 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 99
Number of relapses in the last 12 months prior to screening [Mean (Standard Deviation); unit: relapses/year] | 1.1 (0.59)
Number of relapses in 12 to 24 months prior to screening [Mean (Standard Deviation); unit: relapses/year] | 0.6 (0.80)

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Annualized Relapse Rate (ARR) Based on Confirmed Relapses
Description: A confirmed MS relapse is defined as one accompanied by a clinically-relevant change in the EDSS performed by the Independent EDSS rater, i.e. an increase of at least 0.5 points on the EDSS score, or an increase of 1 point on two functional scores or 2 points on one functional score (excluding changes involving bowel/bladder or cerebral functional system).
  Adjusted ARR was obtained from fitting a negative binomial regression model adjusted for number of relapses in the previous year, baseline number of T1 Gd-enhancing lesions and baseline age as continuous covariates (offset: Natural log of time in study in years).
Time Frame: Baseline up to approximately 12 months
Population: Full analysis set (FAS): comprised of all participants who had signed the Informed Consent and who have had received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: relapses per participant-year
Arm/Group | Ofatumumab
Number analyzed (Participants) | 99
relapses per participant-year | 0.05 [0.02 to 0.13]

2. Other Pre Specified Outcome: Participant Based Annualized Relapse Rate (ARR)
Description: A relapse is an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event which is present for at least 24 hours in the absence of fever or infection.
  A relapse is confirmed by the treating physician when it is accompanied by an increase of at least 0.5 on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
  Participant-based ARR was calculated by taking the total number of relapses observed for a participant divided by the total number of days in study of that participant and multiplied by 365.25.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: relapses per participant-year
Arm/Group | Ofatumumab
Number analyzed (Participants) | 99
relapses per participant-year
  Confirmed relapses | 0.058 (0.2528)
  All relapses | 0.090 (0.3066)

3. Other Pre Specified Outcome: Time Based Annualized Relapse Rate (ARR)
Description: A relapse is an appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event which is present for at least 24 hours in the absence of fever or infection.
  A relapse is confirmed by the treating physician when it is accompanied by an increase of at least 0.5 on the Expanded Disability Status Scale (EDSS) or an increase of 1 point on two different Functional Systems (FS) of the EDSS or 2 points on one of the FS (excluding Bowel/Bladder or Cerebral FS).
  Time-based ARR was calculated by taking the total number of relapses observed for all subjects within an age group divided by the total number of days in study of all subjects within the group and multiplied by 365.25 days.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 1
Measure: Number; unit: relapses per participant-year
Arm/Group | Ofatumumab
Number analyzed (Participants) | 99
relapses per participant-year
  Confirmed relapses | 0.056
  All relapses | 0.089

4. Secondary Outcome: Number of Adverse Events and Serious Adverse Events
Description: Adverse events and SAEs, including clinically significant laboratory data and vital signs which meet the definition of adverse events
Time Frame: Baseline to safety cut-off up to approximately 15.2 months
Population: Safety set (SAF): was identical to FAS in this study. FAS: comprised of all participants who had signed the Informed Consent and who have had received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 99
Participants
  Adverse events (AEs) | 69
  Serious adverse events (SAEs) | 0
  AEs related to treatment | 52
  AEs leading to treatment discontinuation | 0
  AEs leading to treatment interruption | 3

5. Secondary Outcome: Number of Gadolinium (Gd)-Enhancing T1 Lesions Per MRI Scan
Description: Obtained from fitting a negative binomial regression model with log-link function, the total number of Gd-enhancing T1 lesions during the treatment period (per participant) as the response variable. The model includes baseline age and number of Gd-enhancing T1 lesions at baseline as continuous covariates. Natural log of the number of MRI scans is used as the offset.
  MRI scans were performed at screening, month 3 and 12 (end of study) and end of follow up for participants that discontinued treatment. Unscheduled MRIs could be performed at the investigator's judgement.
Time Frame: Baseline up to approximately 12 months
Population: Participants in the Full analysis set (FAS) with available results for this outcome measure. FAS comprised all participants who had signed the Informed Consent and who have had received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: lesions per scan
Arm/Group | Ofatumumab
Number analyzed (Participants) | 98
lesions per scan | 0.04 [0.02 to 0.10]

6. Secondary Outcome: Annualized Rate of New or Enlarging T2 Lesions
Description: Obtained from fitting a negative binomial regression model with log link function, the total number of new or enlarged T2 lesions (relative to baseline/month 3 scan) during the Month 3/treatment period (per participant) as the response variable. Natural log of time from screening scan in years is used as the offset. The model will include baseline age and baseline volume of T2 lesions as continuous covariates.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Lesions per participant-year
Arm/Group | Ofatumumab
Number analyzed (Participants) | 95
Lesions per participant-year
  Relative to baseline | 1.95 [1.38 to 2.75]
  Relative to Month 3 | 0.21 [0.09 to 0.49]

7. Secondary Outcome: Change in T2 Lesion Volume Relative to Baseline
Description: T2 lesion volume as measured by MRI and calculated as post-baseline value - baseline value
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Ofatumumab
Number analyzed (Participants) | 97
milliliters
  Month 3 | -0.03 (1.172)
  Month 12: number analyzed (Participants) | 96
  Month 12 | -0.32 (1.116)

8. Secondary Outcome: Percentage Change in T2 Lesion Volume Relative to Baseline
Description: T2 lesion volume as measured by MRI and percent change calculated as post baseline value - baseline value divided by baseline value multiplied by 100.
Time Frame: Baseline up to approximately 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Ofatumumab
Number analyzed (Participants) | 97
Percent change from baseline
  Month 3 | 1.50 (8.681)
  Month 12: number analyzed (Participants) | 96
  Month 12 | -1.88 (7.083)

ADVERSE EVENTS:
Time Frame: Baseline to end of post treatment follow-up to approximately 18 months
Arm/Group | Ofatumumab
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 69/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab (N=99)
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Asthenia (General disorders and administration site conditions) | 1
Chest discomfort (General disorders and administration site conditions) | 1
Influenza like illness (General disorders and administration site conditions) | 1
Injection site reaction (General disorders and administration site conditions) | 1
Pain (General disorders and administration site conditions) | 1
Pyrexia (General disorders and administration site conditions) | 7
Hepatic function abnormal (Hepatobiliary disorders) | 4
Anaphylactic reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Bacterial infection (Infections and infestations) | 3
COVID-19 (Infections and infestations) | 12
Conjunctivitis (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Groin abscess (Infections and infestations) | 1
Helicobacter infection (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 12
Urinary tract infection (Infections and infestations) | 7
Foot fracture (Injury, poisoning and procedural complications) | 1
Injection related reaction (Injury, poisoning and procedural complications) | 43
Alanine aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Lymphocyte count decreased (Investigations) | 3
Lymphocyte percentage decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Neutrophil percentage increased (Investigations) | 1
White blood cell count decreased (Investigations) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Cervicobrachial syndrome (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Dyssomnia (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT05199571/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT05199571/SAP_001.pdf